CLINICAL TRIAL: NCT05116618
Title: Detection of Resistance Mechanisms in Cerebrospinal Fluid for EGFR-mutant, ALK- and ROS1-rearranged Non-small Cell Lung Cancer Patients With Central Nervous System (CNS) Progression After Evidence of Prior CNS Benefit on Relevant Tyrosine Kinase Inhibitors
Brief Title: Detection of Resistance Mechanisms in Cerebrospinal Fluid for EGFR-mutant, ALK- and ROS1-rearranged
Status: Withdrawn | Type: Observational
Why Stopped: Cancelled by Sponsor
Sponsor: University of Colorado, Denver (Other)
Collaborators: Inivata (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-1193.cc
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Progression; Central Nervous System
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Cohort 1: 10 evaluable enrollments to Cohort 1 with EGFR-mutant NSCLC
  Interventions: Diagnostic Test: InVisionFirst-Lung ctDNA assay
- Cohort 2: 10 evaluable enrollments to Cohort 2 with ALK-rearranged NSCLC
  Interventions: Diagnostic Test: InVisionFirst-Lung ctDNA assay
- Cohort 3: 10 evaluable enrollments to Cohort 3 with ROS1-rearranged NSCLC
  Interventions: Diagnostic Test: InVisionFirst-Lung ctDNA assay

INTERVENTIONS:
Diagnostic Test: InVisionFirst-Lung ctDNA assay — An enhanced tagged/targeted-amplicon sequencing technology for detection of genomic alterations in 36 commonly mutated genes in plasma ctDNA with a sensitivity of 73.9% and specificity of 99.8%.

SUMMARY:
To determine the detection rate of driver oncogenes and resistance mechanisms in cerebrospinal fluid (CSF) for patients with CNS progression (with or without extra-CNS (eCNS) progression) and concordance with plasma/tissue

DETAILED DESCRIPTION:
To determine the detection rate of driver oncogenes and resistance mechanisms in cerebrospinal fluid (CSF) for patients with CNS progression (with or without extra-CNS (eCNS) progression) and concordance with plasma/tissue

* For each individual patient with CNS progression (with or without eCNS progression), compare the molecular status (primary oncogene detection and any mechanisms of identifiable resistance including EGFR-, ALK- and ROS1-mutations, ALK-amplification and bypass-tracks activating mutations) of CSF, plasma and CNS tissue (if data from pathology report is available)
* Molecular status will also be compared with previously obtained and stored plasma/tissue prior to the initiation of current next-generation tyrosine-kinase inhibitor (TKI)

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be aged 18 or older.
4. Pathologically confirmed NSCLC with EGFR-mutation, or ALK- or ROS1-rearrangement and currently on an EGFR, or ALK or ROS1 tyrosine-kinase inhibitor (TKI) as applicable
5. Stage IV NSCLC disease according to AJCC 8th edition
6. Known CNS metastasis prior to current line of therapy with CR/PR/SD for at least 6 months (not purely attributable to prior local therapy such as radiation) on current EGFR, or ALK or ROS1 TKI, confirmed by at least one of the following modalities:

   * CT/MRI for brain metastases
   * characteristic signs and/or symptoms indicating progression,
   * cytology,
   * imaging findings for leptomeningeal disease
7. Confirmed current CNS progression, with or without eCNS progression, on the same TKI based on at least one of the following modalities:

   * CT/MRI for brain metastases
   * characteristic signs and/or symptoms indicating progression,
   * cytology,
   * imaging findings for leptomeningeal disease
8. Prior CNS radiation therapy is allowed

Exclusion Criteria:

1. Has contraindications to receive a lumbar puncture which may include, but are not limited to the following, at the discretion of the patient's oncologist or physician performing the LP:

   * Clinical and/or radiographic evidence of mass effect of raised intracranial pressure (ICP) with risk for cerebral herniation
   * Thrombocytopenia (defined as platelet count ≤ 50 or per local guidelines) or other bleeding diathesis
   * Currently on antiplatelet or anticoagulant therapy at time of consent, for which the thrombosis risk of holding for LP is deemed unacceptable
   * Suspected spinal epidural abscess
   * Any other condition determined by the clinician to be a contraindication
2. History of a second primary malignancy (including a second primary lung cancer) with the exceptions for:

   * Malignancy treated with curative intent and with no known active disease ≥5 years, and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease
3. Women who are documented as pregnant or breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage IV EGFR, ALK, or ROS1-mutant NSCLC who had CNS progression after at least 6 months of stable CNS disease on a relevant TKI are screened. Patients must meet all Inclusion/Exclusion Criteria to participate in the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Determine the detection rate of driver oncogenes and resistance mechanisms in cerebrospinal fluid (CSF) for patients with CNS progression (with or without extra-CNS (eCNS) progression) and concordance with plasma/tissue | 3 years
  * For each individual patient with CNS progression (with or without eCNS progression), compare the molecular status (primary oncogene detection and any mechanisms of identifiable resistance including EGFR-, ALK- and ROS1-mutations, ALK-amplification and bypass-tracks activating mutations) of CSF, plasma and CNS tissue (if data from pathology report is available)
  * Molecular status will also be compared with previously obtained and stored plasma/tissue prior to the initiation of current next-generation tyrosine-kinase inhibitor (TKI)

SECONDARY OUTCOMES:
Compare and contrast mechanisms of resistance in CNS progression versus eCNS progression | 3 years
  * For patients with both CNS and eCNS progression, compare distribution of resistance mechanisms between CSF, plasma, CNS tissue (if data from pathology report is available) and tissue from site of eCNS progression (if data from pathology report is available)
  * Compare distribution of resistance mechanisms in CSF for all patients with CNS progression (with or without eCNS progression) to historical data of distribution of resistance mechanisms to next-generation TKI from ctDNA/tumor tissue samples

OTHER OUTCOMES:
Determine the clinical outcomes of subsequent lines of therapy base on CNS data from this study | 3 years
  ORR in CNS
Determine the clinical outcomes of subsequent lines of therapy base on CNS data from this study | 3 years
  PFS in CNS
Determine the clinical outcomes of subsequent lines of therapy base on eCNS data from this study | 3 years
  ORR in eCNS
Determine the clinical outcomes of subsequent lines of therapy base on eCNS data from this study | 3 years
  PFS in eCNS
Determine the safety of CSF sampling for detection of resistance mechanisms in the context of CNS progression | 3 years
  AEs associated with procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ross Camidge, Principal Investigator — Colorado Research Center
Locations (3):
- United States (3):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Colorado Research Center, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No
whole study will be presented